CLINICAL TRIAL: NCT04195828
Title: Camrelizumab Combined with Apatinib Mesylate Tablets, Nab-paclitaxel and S-1 in the Treatment of Locally Advanced Gastric Cancer: an Multicenter, Open, Randomized, Controlled Clinical Study
Brief Title: Camrelizumab Combined with Apatinib Mesylate Tablets, Nab-paclitaxel and S-1 in the Treatment of Locally Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Arise-FJ-G005
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — camrelizumab; apatinib; 130-nm albumin-bound paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Camrelizumab + Apatinib + nab-paclitaxel +S-1 (Experimental): Camrelizumab combined with Apatinib mesylate tablets, nab-paclitaxel and S-1 in the treatment of locally advanced gastric cancer
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate; Drug: nab-paclitaxel; Drug: S1
- nab-paclitaxel +S-1 (Active Comparator): nab-paclitaxel and S-1 in the treatment of locally advanced gastric cancer
  Interventions: Drug: nab-paclitaxel; Drug: S1

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab One course will last 21 days.Given once every 3 weeks at a dose of 200 mg.
  Arms: Camrelizumab + Apatinib + nab-paclitaxel +S-1
Drug: Apatinib Mesylate — Apatinib One course will last 21 days.Oral administration at a dose of 250 mg everyday。
  Arms: Camrelizumab + Apatinib + nab-paclitaxel +S-1
Drug: nab-paclitaxel — nab-paclitaxel One course will last 21 days。Given twice every 3 weeks at a dose of 125 mg/m2.
Drug: S1 — S-1 was calculated according to body surface area , P.O., bid, d1-d14。And the dosage according body surface area:<1.25m2, 40mg every time;1.25-1.5m2,50mg every time; >1.5m2, 60mg every time

SUMMARY:
To evaluate the clinical efficacy and safety of camrelizumab combined with apatinib mesylate, nab-paclitaxel and S-1

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years of age
* Gastric adenocarcinoma was confirmed by pathology（ including histology or cytology）。
* CT/MRI,PET-CT or laparoscopic exploration were used to confirm the diagnosis of gastric cancer staging as cT2-4a and/or N+ and M0 before operation.
* measurable lesions at least should be detected by CT/MRI examination in accordance with the RECIST1.1.（CT scan of tumor lesion length≥10mm，CT scan short diameter≥15mm，scan slice thicknes 5mm）
* ECOG（Eastern Cooperative Oncology Group）PS（Performance Status）:0-1 scores;
* the expected survival time is more than 12 weeks
* the main organ function is normal, which should meet the following criteria:

  (1) blood routine examination standards should be met（no blood transfusion within 14 days）

  a．HB≥ 100g/L b. WBC≥3×109/L c. ANC≥1.5×109/L d. PLT≥100×109/L （2）biochemical examination shall comply with the following criteria：
  1. BIL<1.5 normal upper limit ULN
  2. ALT and AST<2.5 ULN,GPT≤1.5×ULN
  3. Cr≤1 ULN，CCR（creatinine clearance rate）>60ml/min(Cockcroft-Gault formula)
* women of childbearing age must have a pregnancy test in 7 days before entering the group (in serum), and the results were negative, and willing to use appropriate contraception during the study period and the last 8 weeks after giving drug test; men should have the surgical sterilization, or adopt the appropriate contraceptive methods during the test and the last 8 weeks after giving drug test。
* No other clinical studies were conducted before and during the treatment
* participants is willing to participate in this study, sign the informed consent, have good compliance, cooperate with follow-up.

Exclusion Criteria:

* Previous history of chemotherapy, radiotherapy, targeted drug therapy or immunotherapy
* Patients with contraindications for surgical treatment and chemotherapy or whose physical condition and organ function do not allow for larger abdominal surgery
* patients with metastasis
* Having any active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Patients with vitiligo or cured childhood asthma/allergies who did not need any intervention in adulthood were excluded; Autoimmune hypothyroidism treated with a stable dose of thyroid replacement hormone; Type 1 diabetes with stable doses of insulin
* A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation
* Accompanied by serious heart, lung, liver, kidney disease; Have nerve, mental disease; Jaundice or obstruction of the digestive tract with severe infection
* pregnant or lactating women
* The blood pressure of patients with hypertension cannot be reduced to the normal range by the antihypertensive drugs (systolic pressure >140 mmHg, diastolic pressure >90 mmHg)
* With Ⅰ magnitude of coronary heart disease, arrhythmia (including QTc protracted between male > 450 ms, women > 470 ms) and cardiac insufficiency
* Patients have a clear tendency with gastrointestinal bleeding, including the following situation: local active ulcerative lesions, and fecal occult blood (+ +); with melena and hematemesis history in 2 months; and patients with fecal occult blood (+) and unresected gastric primary tumor; patients with the risk of bleeding should take the gastroscopy test, if it is the gastric cancer, and researchers believe that may results in massive digestive tract hemorrhage；coagulation dysfunction (INR(international normalized ratio)>1.5, APTT(activated partial thromboplastin time)>1.5 ULN), with bleeding tendency;
* Subjects have failed to control good cardiovascular clinical symptoms or disease, including but not limited to: such as: (1) the NYHA class II heart failure (2) above unstable angina pectoris (3) occurred within 1 year (4) have clinical significance of myocardial infarction (mi) room sex or ventricular arrhythmias without clinical intervention on or after clinical intervention is still poorly controlled
* History of interstitial lung disease (except radiation pneumonia without hormone therapy), and history of non-infectious pneumonia
* Patients are positive of urine protein (urine protein detection 2+ or above, or 24 hours urine protein quantitative >1.0g);
* A person who has previously been allergic to any component of camrilizumab or to any component of the drug under study
* The researchers consider those who were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
major pathological response | 4 months
  major pathological response（MPR）

SECONDARY OUTCOMES:
pathological complete response | 4 months
  pathological complete response (pCR)
Objective response rate | 4 months
  Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version. 1.1, and immune-related (ir) RECIST
R0 resection rate | 4 months
  The surgical procedure was total or subtotal gastrectomy with 3 weeks after total neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin JX, Tang YH, Zheng HL, Ye K, Cai JC, Cai LS, Lin W, Xie JW, Wang JB, Lu J, Chen QY, Cao LL, Zheng CH, Li P, Huang CM. Neoadjuvant camrelizumab and apatinib combined with chemotherapy versus chemotherapy alone for locally advanced gastric cancer: a multicenter randomized phase 2 trial. Nat Commun. 2024 Jan 2;15(1):41. doi: 10.1038/s41467-023-44309-5. PMID 38167806